CLINICAL TRIAL: NCT04834609
Title: Identification of Molecular Differences of Adipose-derived Mesenchymal Stem Cells Between Non- Responders and Responders in Treatment of Transsphincteric Perianal Fistulas Using Autologous Fat Graft Injection
Brief Title: Adipose Derived Mesenchymal Stem Cell Characteristics in Anal Fistulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Southern Denmark (Other); UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-MSCs_Anal fistulas
Record Dates: First submitted 2021-03-22; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Perianal Fistula; Adipose Tissue; Tissue Transplantation
Keywords: autologous adipose tissue, mesenchymal stem cells, perianal fistula

STUDY DESIGN:
Masking Description: Characterisation of adipose tissue (AT-MSCs) was performed blinded to the result of the treatment responder/non-responder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection with adipose tissue (Experimental): Injection of freshly collected autologous adipose tissue
  Interventions: Procedure: Injection of autologous adipose tissue in anal fistula

INTERVENTIONS:
Procedure: Injection of autologous adipose tissue in anal fistula

SUMMARY:
This study investigated the cellular and molecular characteristics of AT-MSCs obtained from autologous AT therapy in patients with high transphincteric perianal fistulas of crytoglandular origin. Adipose tissue was injected into anal fistulas. Characteristics of adipose tissue mesenchymal stemcells (AT-MSC) was investigated and compared in patients with fistula that healed after the treatment (responders) to patients who failed to heal (non-responders)

DETAILED DESCRIPTION:
Injection with allogene or autologous stem cells has been reported to be efficient treatment of perianal fistulas. An alternative to this treatment could be injection with freshly collected autologous adipose tissue. In this study 27 patients with cryptoglandular anal fistulas were treated with freshly collected autologous adipose tissue.A clinical assessment of the patient prior to inclusion was undertaken and a loose seton placed for at least 6 weeks prior to fat injection. An MRI of the pelvis was performed before inclusion. Fistulas with secondary tracts and/or cavities were excluded. The operation was performed in one procedure including liposuction and injection of adipose tissue. A sample of adipose tissue from all 27 patients was analyzed. AT-MSCs were isolated and characterized using cellular and molecular analyses. Clinical and MRI-scanning evaluation of fistula healing and evaluation of ano-rectal function was performed after 6 months. AT-MSCs phenotype was compared between responders and non-responders with respect to fistula healing. The evaluation of the AT-MSCs was performed in a blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* high trans-sphincteric fistulas
* fistula confirmed and classified by an MRI.
* seton (> 6 weeks) prior to fat injection
* informed, written consent.

Exclusion Criteria:

Anovaginal fistula

* Active sepsis
* IBD, immunodeficiency, prior pelvic irradiation and malignancy
* Insulin dependent diabetes
* More than 4 prior attempts of fistula closure
* Tobacco smoking or nicotine substitution 8 weeks prior to fat injection.
* Pregnancy
* Psychiatric disorders
* BMI ≥ 35 or BMI<20
* Active tuberculosis
* Patient less than 18 years
* Unable to undergo MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Investigation of cell proliferation of AT-MSCs | At start of treatment
  Cell proliferation of AT-MSCs evaluated as number of cells/per day
Investigation of differentiation potential of AT-MSCs to differentiate into adipocyte | At start of treatment
  Differentiation potential of AT-MSCs: to differentiate into adipocyte measured by Oil-Red O staining and gene expression of adipogenic markers (PPARg and LPL normalized to housekeeping gene beta actin) presented as a Fold change to undifferentiated cells (arbitrary units)
Investigation of differentiation potential of AT-MSCs to differentiate into osteoblast | At start of treatment
  Differentiation potential of AT-MSCs: to differentiate into osteoblast measured by Alizarin S staining and gene expression of osteogenic markers (BGALP and RUNX2 normalized to housekeeping gene beta actin) presented as a Fold change to undifferentiated cells (arbitrary units)
Measurement of gene expression profile of AT-MSCs | At start of treatment
  Gene expression of proinflammatory (NFKB, TNFa, IL1B, IL6) and senescence associated molecules(CDKN2A, TP53, TGFB1, VEGFA, IFNG, IL6) of AT-MSCs in relation to the outcome of fistula treatment (i.e. comparison between responders and non-responders). The data are normalized to housekeeping gene beta actin (arbitrary units)

SECONDARY OUTCOMES:
Healing of anal fistula after treatment | 6 months after last injection of autologous adipose tissue
  Clinical healing defined as closure of the internal and external fistula opening and no discharge evaluated as success rate of the healing in (%)
Evaluation of fistula healing after treatment | 6 months after last injection of autologous adipose tissue
  A combination of Clinical and MRI healing defined as closure of the internal and external fistula opening and no discharge and no fluid filled fistula tracts on evaluated as success rate of the healing in (%)
Functional gastroenterological outcome after treatment | 6 months after last injection of autologous adipose tissue
  Anal continence evaluated as the St. Mark's Score (0-24)
Defecation disorder evaluation after treatment | 6 months after last injection of autologous adipose tissue
  Defecation disorders evaluated as Altomare Obstructed Defecation Score (0-31)
Functional urological outcome after treatment | 6 months after last injection of autologous adipose tissue
  Urinary incontinence evaluated as ICIQ-UI-SF (0-21)

REFERENCES:
- [Derived] Tencerova M, Lundby L, Buntzen S, Norderval S, Hougaard HT, Pedersen BG, Kassem M. Molecular differences of adipose-derived mesenchymal stem cells between non-responders and responders in treatment of transphincteric perianal fistulas. Stem Cell Res Ther. 2021 Nov 24;12(1):586. doi: 10.1186/s13287-021-02644-8. PMID 34819138